CLINICAL TRIAL: NCT00631163
Title: A Multi-Center, Open-label, Non Comparative, Phase II Trial on Efficacy and Safety of ICL670 Given for 1 Year With Dose Adjustments Based on Serum Ferritin in Patients With Chronic Anemia and Transfusional Hemosiderosis Including an Additional 1 Year Extension.
Brief Title: Efficacy and Safety of Deferasirox in Patients With Chronic Anemia and Transfusional Hemosiderosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CICL670A2204; 2006-003337-32 (EudraCT Number); NCT01199003 (obsolete NCT alias)
Record Dates: First submitted 2008-02-27; First posted 2008-03-07 (Estimated); Results first posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Chronic Anemia; Transfusional Hemosiderosis
Keywords: Iron Overload,; Chelation,; MDS,; Chronic Anemia,; Deferasirox,; Transfusional hemosiderosis,
MeSH Terms: conditions — Iron Overload | interventions — Deferasirox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Deferasirox (Experimental): Participants received initial dose of 20 milligrams per kilogram (mg/kg) Deferasirox tablets was administered orally once daily (OD) based on the Participants body weight. The dose of Deferasirox was adjusted to either 10 mg/kg or 30 mg/kg based on the volumes of blood transfusions being administered.
  Interventions: Drug: Deferasirox (ICL670)

INTERVENTIONS:
Drug: Deferasirox (ICL670) — The recommended initial daily dose of Deferasirox is 20 mg/kg body weight.
  Other Names: ICL670

SUMMARY:
The overall purpose of this trial is to further evaluate the efficacy and safety of deferasirox, dosed initially according to the transfusional iron intake, in patients with transfusion dependant anemia related to disorders other than β-thalassemia and sickle cell disease.

During the study, the dose will be adjusted based on serum Ferritin.The overall purpose of the extension is to allow further treatment of patients who have already completed the core study, and to enable collection of long term efficacy and safety data. Patients will continue to receive Deferasirox at the dose they received at the end of the core study.

ELIGIBILITY:
Inclusion criteria (Core):

* Patients with transfusional iron overload due to:
* low or intermediate (INT-1) risk Myelodysplastic Syndrome (MDS)determined via International Prognosis Scoring System (IPSS) criteria
* other congenital or acquired anemias excluding B-thalassemia and sickle cell disease
* Lifetime transfusion history of ≥20 unit (approximately 100 mL/kg) of packed red blood cells or showing evidence of iron overload (serum ferritin >1000 µg/L).
* Able to provide written informed consent
* Life expectancy ≥ 12 months If patient was previously treated with deferiprone, a washout period of one month should occur before the first dose of deferasirox

Inclusion criteria (Extension):

* Patients completing the planned 12-month core study (CICL670A2204).
* Written informed consent obtained from the patient and/or legal guardian on the patient's behalf in accordance with national legislation.

Exclusion criteria (Core and Extension):

* Patients with β-thalassemia, sickle cell disease or myelodysplastic syndrome with an IPSS score being Intermediate-2 or High.
* Patients with serum creatinine > ULN
* Patients with ALT(SGPT) levels > 5 x ULN
* Significant proteinuria as indicated by a urinary protein/creatinine ratio >0.5 mg/mg in a non-first void urine sample on two assessments during the screening period.
* History of HIV positive test result , or of clinical or laboratory evidence of active Hepatitis B or Hepatitis C (HBsAg in the absence of HBsAb OR HCV Ab positive with HCV RNA positive and ALT above the normal range)
* Patients on investigational MDS therapies, including lenalidomide, thalidomide, azacitidine and arsenic trioxide, must have a ≥ 4 week washout period prior to the first dose of study drug.
* Patients with systemic uncontrolled hypertension
* Patients with unstable cardiac disease not controlled by standard medical therapy
* Systemic disease (cardiovascular, renal, hepatic, etc.) which would prevent study treatment
* Pregnancy (as documented in required screening laboratory test) or breast feeding.
* Patients treated with systemic investigational drug within the past 4 weeks or topical investigational drug within the past 7 days
* Other surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of study drug
* Patients being considered by the investigator potentially unreliable and/or not cooperative with regard to the study protocol
* History of hypersensitivity to any of the study drug or excipients
* Sexually active pre-menopausal female patients without adequate contraception. Female patients must use effective contraception or must have undergone clinically documented total hysterectomy and/or oophorectomy, tubal ligation or be postmenopausal defined by amenorrhea for at least 12 months.

Other protocol defined inclusion/exclusion criteria may apply.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2007-10; Primary Completion 2011-01 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Novartis Pharmaceuticals, Study Director — Novartis Pharmeceuticals
Locations (28):
- Japan (20):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Nishinomiya, Hyōgo
  - Novartis Investigative Site, Kahoku-gun, Ishikawa-ken
  - Novartis Investigative Site, Kanazawa, Ishikawa-ken
  - Novartis Investigative Site, Sayama, Osaka
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Shimotsuka-gun, Tochigi
  - Novartis Investigative Site, Simotsuke-city, Tochigi
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Cyuo-ku, Tokyo
  - Novartis Investigative Site, Minato-ku, Tokyo
  - Novartis Investigative Site, Shinagawa-ku, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
  - Novartis Investigative Site, Hiroshima
  - Novartis Investigative Site, Kumamoto
  - Novartis Investigative Site, Kyoto
  - Novartis Investigative Site, Nagasaki
  - Novartis Investigative Site, Toyama
- Novartis Investigative Site, Warsaw, Poland
- Novartis Investigative Site, Singapore, Singapore
- Spain (2):
  - Novartis Investigative Site, Salamanca, Castille and León
  - Novartis Investigative Site, Valencia
- Turkey (Türkiye) (4):
  - Novartis Investigative Site, Adana
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir

REFERENCES:
- [Result] Kohgo Y, Urabe A, Kilinc Y, Agaoglu L, Warzocha K, Miyamura K, Lim LC, Glaser S, Wang C, Wiktor-Jedrzejczak W. Deferasirox Decreases Liver Iron Concentration in Iron-Overloaded Patients with Myelodysplastic Syndromes, Aplastic Anemia and Other Rare Anemias. Acta Haematol. 2015;134(4):233-42. doi: 10.1159/000381893. PMID 26138856
- See also: CICL670A2204 Results at Novartis Clinical Trials Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=2751

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 31 centers and five countries.
Pre-assignment Details: A total of 144 Participants were screened, of which only 102 Participants enrolled in the study. Remaining 42 Participants were considered as screen failures.
Period: Number of Participants in Year 1
Arm/Group | Deferasirox
Started | 102
Completed | 68
Not Completed | 34
Not completed — Adverse Event | 12
Not completed — Withdrawal by Subject | 8
Not completed — Death | 6
Not completed — Lost to Follow-up | 1
Not completed — Patient's condition no longer requires study drug | 1
Not completed — Administrative problems | 6
Period: Number of Participants in Year 2
Arm/Group | Deferasirox
Started | 57
Completed | 52
Not Completed | 5
Not completed — Withdrawal by Subject | 2
Not completed — Adverse Event | 1
Not completed — Protocol Violation | 1
Not completed — Abnormal laboratory value | 1

BASELINE CHARACTERISTICS:
Groups:
- Deferasirox: Participants received initial dose of 20 mg/kg Deferasirox tablets was administered orally OD based on the participants body weight. The dose of Deferasirox was adjusted to either 10 mg/kg or 30 mg/kg based on the volumes of blood transfusions being administered.
Arm/Group | Deferasirox
Number analyzed (Participants) | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (25.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 53
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 46
  Asian | 56
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 53
  Other | 43
  Hispanic or Latino | 4
  Chinese | 2

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Liver Iron Concentration (LIC) to Year 1
Description: Liver iron concentration (LIC), a predictor of iron burden, was measured using relaxation rate magnetic resonance imaging (R2-MRI) technique. Relaxation rate was determined as R2 = 1/relaxation time (T2). The baseline value of LIC of participants was categorized as < 7, ≥ 7 to < 15, and ≥ 15 milligram of iron/tissue dry weight (mg Fe/g dw). A negative change from baseline favored study treatment in reducing LIC.
Time Frame: From the Baseline, Year 1 (End of core study)
Population: The analysis was performed in per-protocol population in core study (PP1 Set), comprising of all enrolled participants who had LIC assessments at baseline and Year 1.
Measure: Mean (Standard Deviation); unit: mg Fe/g dw
Arm/Group | Deferasirox
Number analyzed (Participants) | 50
mg Fe/g dw | -10.9 (11.86)

2. Secondary Outcome: Absolute Change From Baseline in Liver Iron Concentration (LIC) to End of Year 2
Description: Liver Iron Concentration (LIC), a predictor of iron burden, was measured using R2-MRI technique. Relaxation rate was determined as R2 = 1/T2. The baseline value of LIC of participants was categorized as < 7, ≥ 7 to < 15, and ≥ 15 mg Fe/g dw. A negative change from baseline favoured study treatment in reducing LIC.
Time Frame: From the Baseline to End of Year 2 (End of extension study)
Population: The analysis was performed in per-protocol population in core study (PP2 Set), comprising of all enrolled participants who had LIC assessments at baseline and at end of the extension phase.
Measure: Mean (Standard Deviation); unit: mg Fe/g dw
Arm/Group | Deferasirox
Number analyzed (Participants) | 41
mg Fe/g dw | -13.5 (14.10)

3. Secondary Outcome: Absolute Change From Baseline in Liver Iron Concentration (LIC) in Japanese Subgroup
Description: Liver Iron Concentration (LIC), a predictor of iron burden, was measured using R2-MRI technique. Relaxation rate was determined as R2 = 1/T2. The baseline value of LIC was < 7, ≥ 7 to < 15, and ≥ 15 mg Fe/g dw. A negative change from baseline favoured study treatment in reducing LIC.
Time Frame: From the Baseline, End of Year 1 (End of core study), End of Year 2 (End of extension study)
Population: The analysis was performed in PP1 set in Japanese subgroup defined as all participants who were enrolled in Japan for core study (Year 1) and PP2 set in Japanese subgroup for extension study (Year 2). Here, 'n' signifies the participants reviewed for Liver Iron Concentration (LIC) in Japanese subgroup for each group, respectively.
Measure: Mean (Standard Deviation); unit: mg Fe/g dw
Arm/Group | Deferasirox
Number analyzed (Participants) | 57
mg Fe/g dw
  Year 1: number analyzed (Participants) | 31
  Year 1 | -13.9 (10.21)
  Year 2: number analyzed (Participants) | 26
  Year 2 | -18.4 (12.48)

4. Secondary Outcome: Absolute Change From Baseline in Serum Ferritin Levels to Year 2
Description: Serum ferritin was a marker for the monitoring of chelation therapy. Ferritin protein stores iron and provides overall iron levels, higher ferritin in blood showed more iron content.
Time Frame: From the Baseline up to Year 2 (End of extension study)
Population: The analysis was performed in PP2 Set population and Japanese subgroup. Here, "Number of subjects analyzed" signifies the participants assessed for serum ferritin during the study for each arm, respectively.
Measure: Mean (Standard Deviation); unit: nanogram(s)/millilitre
Groups:
- All Randomized Participants; Japanese Participants: Participants received initial dose of 20 mg/kg Deferasirox tablets was administered orally OD based on the Participants body weight. The dose of Deferasirox was adjusted to either 10 mg/kg or 30 mg/kg based on the volumes of blood transfusions being administered.
Arm/Group | All Randomized Participants | Japanese Participants
Number analyzed (Participants) | 102 | 53
nanogram(s)/millilitre | -677.9 (4462.11) | -892.8 (5724.89)

5. Secondary Outcome: Absolute Serum Ferritin Levels Over 2 Years
Description: as for outcome 4
Time Frame: From the Baseline, Year 1 (End of core study), Year 2 (End of extension study)
Population: The analysis was performed in PP1 set population for core study (Year 1) and PP2 set population for extension study (Year 2) and Japanese subgroup. Here, "Number of participants analysed" signifies the subjects assessed for serum ferritin during the study for each arm, respectively.
Measure: Mean (Standard Deviation); unit: nanogram(s)/millilitre
Arm/Group | All Randomized Participants | Japanese Participants
Number analyzed (Participants) | 50 | 31
nanogram(s)/millilitre
  Year 1 | 2653.3 (2952.07) | 2903.5 (3376.00)
  Year 2 | 2092.4 (2287.11) | 2114.8 (2391.31)

6. Secondary Outcome: Total Body Iron Elimination Rate (TBIE), Iron Intake, Iron Excretion/Iron Intake and Chelation Efficiency After 2 Years
Description: Total body iron excretion (TBIE)was used to investigate the chelation efficacy of Deferasirox therapy. TBIE rate was estimated based on the iron influx as determined by the amount of red cells transfused and the change in total body iron (TBI) stores.
Time Frame: From the Baseline, Year 2 (End of extension study)
Population: The analysis was performed in PP2 set population and Japanese/tim subgroup. Here, "Number of participants analyzed" included all participants who were evaluable for the specified categories.
Measure: Mean (Standard Deviation); unit: mg/kg/day
Groups:
- Deferasirox (Extension Study); Japanese Participants: Participants received initial dose of 20 mg/kg Deferasirox tablets was administered orally OD based on the Participants body weight. The dose of Deferasirox was adjusted to either 10 mg/kg or 30 mg/kg based on the volumes of blood transfusions being administered.
Arm/Group | Deferasirox (Extension Study) | Japanese Participants
Number analyzed (Participants) | 41 | 26
mg/kg/day
  TBIE | 0.46 (0.252) | 0.54 (0.215)
  Iron intake: number analyzed (Participants) | 40 | 26
  Iron intake | 0.27 (0.150) | 0.27 (0.160)
  Iron excretion/iron intake: number analyzed (Participants) | 40 | 26
  Iron excretion/iron intake | 2.00 (1.368) | 2.44 (1.417)
  Chelation efficiency | 0.40 (0.221) | 0.50 (0.177)

7. Secondary Outcome: Correlation of LIC and Serum Ferritin at Core and Extension Study
Description: LIC, a predictor of iron burden, was measured using R2-MRI technique. Relaxation rate was determined as R2 = 1/T2. The baseline value of LIC was < 7, ≥ 7 to < 15, and ≥ 15 mg Fe/g dw. Serum ferritin was a marker for the monitoring of chelation therapy. Ferritin protein stores iron and provides overall iron levels, higher ferritin in blood showed more iron content. The correlation between absolute change in LIC and absolute change in serum ferritin was determined.
Time Frame: From the Baseline, Year 1 (End of core study), Year 2 (End of extension study)
Population: The analysis was performed in PP1 set for core study (Year 1) and PP2 set for extension study (Year 2). Here, "Number of subjects analysed" signifies the subjects assessed for LIC and serum ferritin during the study for each arm, respectively.
Measure: Number; unit: Correlation coefficient
Groups:
- Deferasirox (Core Study); Deferasirox (Extension Study): Participants received initial dose of 20 mg/kg Deferasirox tablets was administered orally OD based on the Participants body weight. The dose of Deferasirox was adjusted to either 10 mg/kg or 30 mg/kg based on the volumes of blood transfusions being administered.
Arm/Group | Deferasirox (Core Study) | Deferasirox (Extension Study)
Number analyzed (Participants) | 50 | 40
Correlation coefficient | 0.291 | 0.325

8. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), Adverse Event of Special Interest (AESI), Discontinuation and Interruption
Description: Adverse events (AEs) were defined as any unfavorable and unintended diagnosis, symptom, sign (including an abnormal laboratory finding), syndrome or disease which either occurs during study, having been absent at baseline, or, if present at baseline, appears to worsen. Serious adverse events (SAEs) were defined as any untoward medical occurrences that result in death, are life threatening, require hospitalisation, cause persistent or significant disability/incapacity, result in congenital anomalies or birth defects, or are other conditions which in judgement of investigators represent significant hazards. Death was defined as a fatal event leading to permanent cessation of all vital functions of the body.
Time Frame: From the Baseline up to Year 2 (End of extension study)
Population: The analysis was performed in the safety set (SAF) population, defined as subjects who received at least one dose of study drug, which was defined as at least one administration record with a valid date and an actual total daily dose administrated above zero, and Japanese sub-group.
Measure: Number; unit: participants
Arm/Group | All Randomized Participants
Number analyzed (Participants) | 102
participants
  Adverse Events | 97
  Serious Adverse Events (SAE) | 46
  Serious Adverse Events (SAE) with suspected relationship to study drug | 10
  Death | 6
  Adverse event leading to discontinuation of study drug | 14
  Adverse event leading to dose adjustment/interruption | 67
  Adverse Event of Special Interest (AESI) | 62
  Adverse Event With Suspected Relationship to Study drug | 65

9. Secondary Outcome: Number of Participants With Clinically Significant Ophthalmological Abnormalities
Description: Clinically significant changes in left eye and right eye were assessed by the investigator based on methods like visual acuity, slit lamp examination, tonometry and fundus oculi.
Time Frame: At 2 years (End of extension study)
Population: The analysis was performed in the SAF population, defined as subjects who received at least one dose of study drug, which was defined as at least one administration. These participants comprise 2 year completer groups
Measure: Number; unit: participants
Arm/Group | All Randomized Participants
Number analyzed (Participants) | 50
participants
  Normal | 24
  Abnormal, Clinically Insignificant | 14
  Abnormal, Clinically Significant | 9
  Not Available | 3
  Total | 50

ADVERSE EVENTS:
Time Frame: From the Baseline up to Year 2 (End of extension study)
Description: The analysis was performed on safety set population defined as all participants who received study drug and had at least one post-baseline safety assessment.
Groups:
- Myelodysplastic Syndrome: A group of disorders caused when something disrupts the production of blood cells.
- Aplastic Anemia: Aplastic anemia is a condition that occurs when your body stops producing enough new blood cells. The condition leaves you fatigued and more prone to infections and uncontrolled bleeding.
- Other: Very rare diseases (e.g. Diamond Blackfan anemia, myelofibrosis, specific enzyme deficiency).
Arm/Group | Myelodysplastic Syndrome | Aplastic Anemia | Other
All-Cause Mortality (participants affected / at risk) | 2/42 | 3/29 | 1/31
Serious Adverse Events (participants affected / at risk) | 22/42 | 14/29 | 10/31
Other Adverse Events (participants affected / at risk) | 39/42 | 25/29 | 25/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Myelodysplastic Syndrome (N=42) | Aplastic Anemia (N=29) | Other (N=31)
ANAEMIA (Blood and lymphatic system disorders) | 1 | 0 | 1
APLASTIC ANAEMIA (Blood and lymphatic system disorders) | 0 | 3 | 0
DISSEMINATED INTRAVASCULAR COAGULATION (Blood and lymphatic system disorders) | 2 | 1 | 0
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 2 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 2 | 0 | 0
ATRIAL FLUTTER (Cardiac disorders) | 1 | 0 | 0
CARDIAC FAILURE (Cardiac disorders) | 1 | 0 | 0
PERICARDITIS (Cardiac disorders) | 1 | 0 | 0
DELAYED PUBERTY (Endocrine disorders) | 0 | 0 | 1
CATARACT (Eye disorders) | 0 | 0 | 1
RETINAL HAEMORRHAGE (Eye disorders) | 0 | 0 | 1
ASCITES (Gastrointestinal disorders) | 1 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 0 | 0 | 1
ENTEROCOLITIS (Gastrointestinal disorders) | 1 | 0 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 2 | 0
GASTROINTESTINAL ULCER (Gastrointestinal disorders) | 1 | 0 | 0
PERIODONTAL DISEASE (Gastrointestinal disorders) | 1 | 0 | 0
PERIODONTITIS (Gastrointestinal disorders) | 1 | 0 | 0
RADICULAR CYST (Gastrointestinal disorders) | 1 | 0 | 0
VOMITING (Gastrointestinal disorders) | 0 | 0 | 1
CHEST DISCOMFORT (General disorders) | 1 | 0 | 0
DISUSE SYNDROME (General disorders) | 1 | 0 | 0
FATIGUE (General disorders) | 1 | 0 | 0
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 1 | 0 | 0
GENERALISED OEDEMA (General disorders) | 1 | 0 | 0
MALAISE (General disorders) | 0 | 0 | 1
MULTI-ORGAN FAILURE (General disorders) | 2 | 0 | 0
PYREXIA (General disorders) | 6 | 2 | 1
CHOLECYSTITIS (Hepatobiliary disorders) | 1 | 0 | 0
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 1 | 0 | 0
HYPERSENSITIVITY (Immune system disorders) | 0 | 2 | 0
BACTERIAL INFECTION (Infections and infestations) | 1 | 0 | 0
BRONCHITIS (Infections and infestations) | 1 | 0 | 0
BRONCHOPNEUMONIA (Infections and infestations) | 1 | 1 | 0
CELLULITIS (Infections and infestations) | 0 | 0 | 1
ENTEROCOLITIS INFECTIOUS (Infections and infestations) | 1 | 0 | 0
FUNGAEMIA (Infections and infestations) | 1 | 0 | 0
FUNGAL OESOPHAGITIS (Infections and infestations) | 1 | 0 | 0
GASTRITIS VIRAL (Infections and infestations) | 1 | 0 | 0
GASTROENTERITIS (Infections and infestations) | 0 | 1 | 1
HERPES ZOSTER (Infections and infestations) | 1 | 1 | 0
INFECTION (Infections and infestations) | 1 | 0 | 0
INFLUENZA (Infections and infestations) | 0 | 1 | 0
MENINGITIS (Infections and infestations) | 0 | 1 | 0
ORAL HERPES (Infections and infestations) | 1 | 0 | 0
PARONYCHIA (Infections and infestations) | 0 | 1 | 0
PERTUSSIS (Infections and infestations) | 0 | 0 | 1
PHARYNGITIS (Infections and infestations) | 1 | 0 | 0
PNEUMONIA (Infections and infestations) | 4 | 3 | 0
SEPSIS (Infections and infestations) | 2 | 1 | 0
SEPTIC SHOCK (Infections and infestations) | 2 | 0 | 0
URINARY TRACT INFECTION (Infections and infestations) | 3 | 0 | 0
VIRAL INFECTION (Infections and infestations) | 0 | 0 | 1
ZYGOMYCOSIS (Infections and infestations) | 0 | 0 | 1
CONTUSION (Injury, poisoning and procedural complications) | 0 | 1 | 0
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
TOOTH FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
TRAUMATIC HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 | 1 | 0
TRAUMATIC INTRACRANIAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 | 1 | 0
BODY HEIGHT BELOW NORMAL (Investigations) | 0 | 0 | 1
C-REACTIVE PROTEIN INCREASED (Investigations) | 0 | 1 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 0 | 0
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 2 | 0 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
BONE SWELLING (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
ABDOMINAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
BLADDER NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
MYELODYSPLASTIC SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
MYELOFIBROSIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
RECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
CEREBELLAR HAEMORRHAGE (Nervous system disorders) | 0 | 1 | 0
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 0 | 1 | 0
CEREBRAL INFARCTION (Nervous system disorders) | 0 | 1 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 | 0 | 0
DIZZINESS (Nervous system disorders) | 1 | 0 | 0
NEUROSIS (Psychiatric disorders) | 0 | 0 | 1
FANCONI SYNDROME ACQUIRED (Renal and urinary disorders) | 0 | 0 | 1
NEPHROLITHIASIS (Renal and urinary disorders) | 1 | 0 | 0
ADENOIDAL HYPERTROPHY (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
HAEMORRHAGE SUBCUTANEOUS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
PANNICULITIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
URTICARIA (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Myelodysplastic Syndrome (N=42) | Aplastic Anemia (N=29) | Other (N=31)
ANAEMIA (Blood and lymphatic system disorders) | 5 | 1 | 1
APLASTIC ANAEMIA (Blood and lymphatic system disorders) | 0 | 2 | 0
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 2 | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 3 | 2 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 4 | 2 | 0
CARDIAC FAILURE (Cardiac disorders) | 4 | 2 | 1
TACHYCARDIA (Cardiac disorders) | 3 | 2 | 1
CATARACT (Eye disorders) | 4 | 2 | 0
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 3 | 1 | 0
EYE PAIN (Eye disorders) | 1 | 2 | 0
RETINAL HAEMORRHAGE (Eye disorders) | 2 | 3 | 3
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 0 | 3 | 1
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 3 | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 7 | 4 | 2
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2 | 3 | 1
APHTHOUS STOMATITIS (Gastrointestinal disorders) | 1 | 2 | 1
CONSTIPATION (Gastrointestinal disorders) | 13 | 5 | 3
DENTAL CARIES (Gastrointestinal disorders) | 3 | 2 | 0
DIARRHOEA (Gastrointestinal disorders) | 10 | 7 | 5
GASTRITIS (Gastrointestinal disorders) | 1 | 2 | 0
HAEMORRHOIDS (Gastrointestinal disorders) | 3 | 3 | 0
NAUSEA (Gastrointestinal disorders) | 9 | 6 | 2
STOMATITIS (Gastrointestinal disorders) | 8 | 7 | 0
VOMITING (Gastrointestinal disorders) | 3 | 4 | 0
ASTHENIA (General disorders) | 2 | 2 | 1
CHEST PAIN (General disorders) | 1 | 3 | 0
FACE OEDEMA (General disorders) | 2 | 2 | 0
FATIGUE (General disorders) | 2 | 1 | 3
MALAISE (General disorders) | 2 | 4 | 2
OEDEMA PERIPHERAL (General disorders) | 14 | 7 | 1
PYREXIA (General disorders) | 11 | 9 | 6
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 2 | 2 | 0
BRONCHITIS (Infections and infestations) | 2 | 0 | 4
CYSTITIS (Infections and infestations) | 5 | 3 | 0
EAR INFECTION (Infections and infestations) | 0 | 0 | 2
FURUNCLE (Infections and infestations) | 0 | 2 | 0
HERPES SIMPLEX (Infections and infestations) | 3 | 0 | 0
HERPES ZOSTER (Infections and infestations) | 4 | 0 | 0
INFLUENZA (Infections and infestations) | 1 | 3 | 2
NASOPHARYNGITIS (Infections and infestations) | 14 | 10 | 6
ORAL CANDIDIASIS (Infections and infestations) | 3 | 0 | 0
OTITIS MEDIA (Infections and infestations) | 0 | 2 | 1
OTITIS MEDIA CHRONIC (Infections and infestations) | 0 | 2 | 0
PHARYNGITIS (Infections and infestations) | 3 | 1 | 2
TONSILLITIS (Infections and infestations) | 2 | 0 | 3
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 2 | 9
URINARY TRACT INFECTION (Infections and infestations) | 3 | 0 | 3
ALLERGIC TRANSFUSION REACTION (Injury, poisoning and procedural complications) | 3 | 1 | 1
CONTUSION (Injury, poisoning and procedural complications) | 6 | 3 | 0
FALL (Injury, poisoning and procedural complications) | 2 | 3 | 0
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1 | 2 | 0
TOOTH INJURY (Injury, poisoning and procedural complications) | 0 | 2 | 0
TRANSFUSION REACTION (Injury, poisoning and procedural complications) | 4 | 2 | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 3 | 1 | 3
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 2 | 1
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 1 | 3 | 2
BLOOD CREATININE INCREASED (Investigations) | 16 | 8 | 2
C-REACTIVE PROTEIN INCREASED (Investigations) | 4 | 5 | 0
PROTEIN URINE PRESENT (Investigations) | 3 | 1 | 5
WEIGHT DECREASED (Investigations) | 2 | 2 | 2
DECREASED APPETITE (Metabolism and nutrition disorders) | 7 | 4 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 5 | 3 | 0
DIABETES MELLITUS (Metabolism and nutrition disorders) | 4 | 2 | 1
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 4 | 4 | 1
HYPOKALAEMIA (Metabolism and nutrition disorders) | 3 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 7 | 2 | 1
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 3 | 3 | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 3 | 1 | 3
MYALGIA (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 5 | 2 | 3
MYELODYSPLASTIC SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1 | 0
DYSGEUSIA (Nervous system disorders) | 1 | 2 | 0
HEADACHE (Nervous system disorders) | 8 | 4 | 3
SOMNOLENCE (Nervous system disorders) | 1 | 2 | 1
DELIRIUM (Psychiatric disorders) | 3 | 0 | 0
INSOMNIA (Psychiatric disorders) | 6 | 1 | 1
PROTEINURIA (Renal and urinary disorders) | 4 | 1 | 1
RENAL FAILURE (Renal and urinary disorders) | 4 | 3 | 2
RENAL IMPAIRMENT (Renal and urinary disorders) | 4 | 6 | 2
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 5
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 | 3 | 4
MADAROSIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
PETECHIAE (Skin and subcutaneous tissue disorders) | 3 | 0 | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 2 | 4 | 1
RASH (Skin and subcutaneous tissue disorders) | 11 | 3 | 1
SKIN ULCER (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
HYPOTENSION (Vascular disorders) | 2 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes